CLINICAL TRIAL: NCT04196036
Title: Cumulative Pregnancy Rates and Direct Healthcare Cost Analysis of Two Different Strategies: Fresh Cleavage-stage Embryo Transfer (ET) on Day 3 With Vitrification of Supernumerary Embryos on Day 3 Versus Day 5
Brief Title: Day 3 Fresh Transfer Followed by Day 3 or Day 5 Vitrification of Supernumerary Embryos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sophie Debrock (Other)
Responsible Party: Sponsor-Investigator, Sophie Debrock, Professor, PhD, KU Leuven
Organization: KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S60974
Record Dates: First submitted 2018-01-15; First posted 2019-12-12 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Subfertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day 3 vitrification (Active Comparator): Day of vitrification of supernumerary embryos is day 3
  Interventions: Procedure: Day of vitrification
- Day 5 vitrification (Active Comparator): Day of vitrification of supernumerary embryos is day5
  Interventions: Procedure: Day of vitrification

INTERVENTIONS:
Procedure: Day of vitrification — Supernumerary embryos after fresh transfer on Day 3 after oocyte aspiration are either vitrified on Day 3 or are kept in culture until Day 5 and vitrified on Day 5

SUMMARY:
This monocenter academic study aims to evaluate the effectiveness and cost effectiveness of two different strategies: fresh Embryo Transfer (ET) on day 3 followed by cryopreservation of cleavage-stage (Day 3) embryos versus blastocyst-stage (Day 5) embryos.

The primary outcome is the cumulative pregnancy rate after all transfers (fresh and/or frozen embryo transfer cycles which might take about 1 year), up to two sequential cycles. The secondary outcome concerns a cost analysis of both strategies from the healthcare payer's perspective.

ELIGIBILITY:
Inclusion Criteria:

* subfertile women planned for the first or second oocyte retrieval for in vitro fertilisation (IVF)/Intracytoplasmic sperm injection (ICSI) treatment
* who are older than 18 and less than 38 years old
* who have normal Follicle Stimulating Hormone (FSH) and normal Anti-Mullerian Hormone (AMH) levels

Exclusion Criteria:

* treatment with donor oocytes or donor embryos
* patients planned for Pre-implantation Genetic Diagnosis (PGD)
* Patients with BMI>30
* patients with endometriosis grade III-IV

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
cumulative pregnancy rate | Cumulative pregnancy is measured after two consecutive IVF cycles including fresh and frozen transfers which might take about 1 year
  The cumulative pregnancy rate after all transfers (fresh and/or frozen embryo transfer cycles)

SECONDARY OUTCOMES:
cost analysis | Cumulative pregnancy is measured after two consecutive IVF cycles including fresh and frozen transfers which might take about 1 year
  cost analysis of day 3 and day 5 vitrification strategy

CONTACTS AND LOCATIONS:
Locations (1):
- Leuven University Fertility Center, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mengels A, Van Muylder A, Peeraer K, Luyten J, Laenen A, Spiessens C, Debrock S. Cumulative pregnancy rates of two strategies: Day 3 fresh embryo transfer followed by Day 3 or Day 5/6 vitrification and embryo transfer: a randomized controlled trial. Hum Reprod. 2024 Jan 5;39(1):62-73. doi: 10.1093/humrep/dead222. PMID 37886820